CLINICAL TRIAL: NCT00430053
Title: Pathogenesis And Course Of Cutaneous T-Cell Lymphoma
Brief Title: Clinical Evaluations and Laboratory Studies to Study the Disease Course in Patients With Cutaneous T-Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: 040081; 04-C-0081; CDR0000354510; NCT00075322 (obsolete NCT alias)
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Lymphoma
Keywords: stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Gene Rearrangement; Polymerase Chain Reaction; Flow Cytometry; Immunohistochemistry; Biopsy

INTERVENTIONS:
Genetic: gene rearrangement analysis
Genetic: polymerase chain reaction
Genetic: proteomic profiling
Other: flow cytometry
Other: immunohistochemistry staining method
Procedure: biopsy

SUMMARY:
RATIONALE: Gathering information about patients with cutaneous T-cell lymphoma over time may help doctors learn more about the disease.

PURPOSE: This natural history study is collecting disease-related health information over time from patients with cutaneous T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Follow the disease course of patients with cutaneous T-cell lymphoma.
* Provide a patient population for study by proteomic and molecular analysis.
* Develop a mechanism for screening by a Tumor Board for enrollment of patients in therapeutic clinical trials.

Secondary

* Develop a tissue bank for future disease study using specimens from these patients.
* Provide community outreach by offering a second opinion regarding treatment of this disease in these patients and, in limited cases, provide standard-of-care treatment to these patients.
* Develop an algorithm for screening and evaluating this disease in these patients.

OUTLINE: Patients undergo disease assessment by physical examination, full-body photographic documentation of skin disease, biopsy, and blood sampling at baseline and then at least annually thereafter. Proteomic and molecular methods are used to analyze samples. Biopsies may be examined using histologic and immunohistochemical methods. Blood may be analyzed by polymerase chain reaction for clonal T-cell gene rearrangements or by flow cytometry.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Histologically confirmed stage IA-IVB cutaneous T-cell lymphoma (CTCL) (mycosis fungoides or Sézary syndrome)
  * Other histologically and clinically confirmed primary or secondary CTCL
  * Histologically and clinically confirmed pre-CTCL skin condition, including large plaque parapsoriasis and lymphomatoid papulosis
* Measurable disease by skin lesion assessment or Sézary cell count

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Human T-cell lymphotrophic virus (HTLV) I/II negative
* Not pregnant
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-01; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Disease course of patients with cutaneous T-cell lymphoma (CTCL)
Provide a patient population for study by proteomic and molecular analysis
Mechanism for screening by a Tumor Board for enrollment of patients in therapeutic clinical trials

SECONDARY OUTCOMES:
Develop a tissue bank for future disease study
Offer a second opinion regarding treatment of CTCL and, in limited cases, provide standard-of-care treatment
Develop an algorithm for screening and evaluating CTCL

CONTACTS AND LOCATIONS:
Overall Officials: Mark C. Udey, MD, PhD, Principal Investigator — NCI - Dermatology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States